CLINICAL TRIAL: NCT02175862
Title: Long-term Evaluation of Patients Treated by an Emergency Medical Helicopter
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Kamilia S. Funder, MD., Rigshospitalet, Denmark
Other Study IDs: ALH1-KF-2014
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Wounds and Injuries
Keywords: Helicopter Emergency Medical Service; Trauma; Early retirement; ISS; Quality of life
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Trauma patients before PS-HEMS: The "before" period was between december 1 2009 to april 30 2010 (five months).
- Traume patients after PS-HEMS: The "after" period was between may 1 2010 to april 30 2011 (12 months).

SUMMARY:
In May 2010 the first danish physician-staffed Helicopter Emergency Medical Service (PS-HEMS) was implemented in Region Zealand and the Capital Region (excluding Bornholm) of Denmark.

In relation to the introduction of PS-HEMS, a team of collaborators lead by Rasmus Hesselfeldt, conducted an observational study to investigate the possible effects on time to definitive care, secondary transfers and 30-day mortality in a "before" and "after" design.

Results showed reduced time from first dispatch to arrival at the trauma centre from 218 min to 90 min. Secondary transfers to the trauma centre dropped from 50 % to 34 % and 30-day mortality significantly reduced from 29 % to 14 % in the year after implementation.

The present study is an observational cohort study with long-term follow-up of the same trauma population as mentioned above. Patients were followed until may 1st, 2014.

Primary outcome is early retirement and secondary outcomes are quality of life and mortality.

The investigators hypothesize that a greater proportion of trauma patients in the "after" period will remain in occupation after approx. 3 to 4.5 years compared with trauma patients treated in the "before" period.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated by a trauma team in the catchment area of PS-HEMS.

For all labor market attachment analysis the investigators only include patients between 18 to 60 years of age. For all other analysis (mortality and quality of life) there are no age limits.

Exclusion Criteria:

* Patients transported by private means or by the police.
* Patients who at the emergency department were categorized as non-trauma patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All trauma patients treated in the catchment area of PS-HEMS in a 17-month period from 1 December 2009 to 30 April 2011 (1791 patients).
Sampling Method: Probability Sample
Enrollment: 1791 (Actual)
Dates: Start 2009-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Labor market attachment | 3 - 4.5 years after trauma
  Primary analysis: Risk of early retirement Secondary analysis: Risk of reduced work capability

SECONDARY OUTCOMES:
Health-related quality of life | 3 - 4.5 years after trauma
  Health-related quality of life is measured using the Danish version of the Short Form 36 (SF-36) questionaire.
All cause mortality | 3 - 4.5 years after trauma
  Primary analysis: Risk of death. Secondary analysis: Predictors of death

CONTACTS AND LOCATIONS:
Overall Officials: Kamilia S. Funder, MD, Principal Investigator — Department of Anesthesia, Center of Head and Orthopedics, section 4231, Copenhagen University Hospital, Rigshospitalet; Jacob Steinmetz, MD, PhD, Study Director — Trauma Center, Copenhagen University Hospital, Rigshospitalet
Locations (1):
- Department Of Anesthesia, Center of Head and Orthopedics, section 4231, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Kuhlman MB, Lohse N, Sorensen AM, Larsen CF, Christensen KB, Steinmetz J. Impact of the severity of trauma on early retirement. Injury. 2014 Mar;45(3):618-23. doi: 10.1016/j.injury.2013.09.007. Epub 2013 Sep 16. PMID 24176678
- [Background] Hesselfeldt R, Steinmetz J, Jans H, Jacobsson ML, Andersen DL, Buggeskov K, Kowalski M, Praest M, Ollgaard L, Hoiby P, Rasmussen LS. Impact of a physician-staffed helicopter on a regional trauma system: a prospective, controlled, observational study. Acta Anaesthesiol Scand. 2013 May;57(5):660-8. doi: 10.1111/aas.12052. Epub 2013 Jan 7. PMID 23289798
- [Background] Overgaard M, Hoyer CB, Christensen EF. Long-term survival and health-related quality of life 6 to 9 years after trauma. J Trauma. 2011 Aug;71(2):435-41. doi: 10.1097/TA.0b013e31820e7ec3. PMID 21427614
- [Background] Ringburg AN, Polinder S, Meulman TJ, Steyerberg EW, van Lieshout EM, Patka P, van Beeck EF, Schipper IB. Cost-effectiveness and quality-of-life analysis of physician-staffed helicopter emergency medical services. Br J Surg. 2009 Nov;96(11):1365-70. doi: 10.1002/bjs.6720. PMID 19847879
- [Background] MacKenzie EJ, Shapiro S, Smith RT, Siegel JH, Moody M, Pitt A. Factors influencing return to work following hospitalization for traumatic injury. Am J Public Health. 1987 Mar;77(3):329-34. doi: 10.2105/ajph.77.3.329. PMID 3812840
- [Background] Baker SP, O'Neill B, Haddon W Jr, Long WB. The injury severity score: a method for describing patients with multiple injuries and evaluating emergency care. J Trauma. 1974 Mar;14(3):187-96. No abstract available. PMID 4814394
- [Background] Bjorner JB, Damsgaard MT, Watt T, Groenvold M. Tests of data quality, scaling assumptions, and reliability of the Danish SF-36. J Clin Epidemiol. 1998 Nov;51(11):1001-11. doi: 10.1016/s0895-4356(98)00092-4. PMID 9817118